CLINICAL TRIAL: NCT06130904
Title: Effect of Academic Detailing on Opioid Prescribing by Dentists to Adolescents and Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: The Benter Foundation (Unknown)
Responsible Party: Principal Investigator, Chad Brummett, Professor of Anesthesiology Research, Senior Associate Chair for Research, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HUM00238416
Record Dates: First submitted 2023-11-08; First posted 2023-11-14 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Opioid Prescribing
Keywords: Dentist; Oral and maxillofacial surgeon

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The analysts will be blinded using codes to prevent bias in analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Academic detailing intervention (Experimental)
  Interventions: Behavioral: Academic detailing
- Control group (No Intervention): Control dentists will receive no intervention at all. Only dentist's prescribing data will be analyzed.

INTERVENTIONS:
Behavioral: Academic detailing — Eligible dentists/oral surgeons will have one visit (30 minutes or less) at the dentist's office. During the initial visit, the detailers will discuss the evidence against routine opioid prescribing to adolescents and young adults for most common surgeries performed by dentists and oral surgeons, the harms of dental opioid exposure in adolescents and young adults, and the benefits and feasibility of relying on non-opioids as a first line option for routine dental procedures among adolescents and young adults. A survey will be completed to assess the satisfaction regarding the intervention. A professionally designed packet of information on reducing use of opioids for routine procedures will also be given.
  There may also be a second optional follow-up visit conducted virtually for any participants that wish to discuss further with the detailer. The second visit may occur any time between the initial visit and March 31, 2024.
  Arms: Academic detailing intervention

SUMMARY:
This randomized controlled trial will test whether an academic detailing educational outreach intervention (referred to as "academic detailing" throughout) decreases opioid prescribing to patients aged 13-30 years among high-prescribing dentists in Southeast Michigan. The primary objective is to evaluate whether an academic detailing intervention reduces the number of dispensed opioid prescriptions to patients aged 13-30 years.

DETAILED DESCRIPTION:
Using 2023 IQVIA Longitudinal Prescription Database, the study team will identify dentists in the 85th-94th percentile of dispensed opioid prescriptions to patients aged 13-30 years from January 1, 2023 through September 30, 2023 and practice in high-population counties in Southeast Michigan. The study team will randomize these dentists into two study arms. Dentists in the intervention arm will receive an academic detailing session focused on evidence-based pain management education. Dentists in the control will not receive any intervention and will not be contacted. Prescribing will be evaluated using IQVIA data for differential change in the number of dispensed opioid prescriptions to patients aged 13-30 years between the 8 months before and the 8 months after the academic detailing intervention period among intervention versus control dentists.

ELIGIBILITY:
Inclusion Criteria for the practioners:

* General dentist, dental subspecialist, or oral and maxillofacial surgeon practicing in the State of Michigan that accounted for at least one dispensed opioid prescription to patients aged 13-30 years during January 1, 2023 through September 30, 2023.

Exclusion Criteria for the practioners:

* Dentist is not included in the OneKey database
* Dentist has an address in OneKey that corresponds to an academic institution (thus excluding residents/fellows and attendings at academic institutions)
* Dentist did not practice in a high-population county in Southeast Michigan, such as Wayne, Oakland, Macomb, Washtenaw, Ingham, Genesee, during the pre-intervention period (April 1, 2023 through November 30, 2023).
* Dentist was not in the 85th-94th percentile of dispensed opioid prescriptions to patients aged 13-30 years during January 1, 2023 through September 30, 2023.
* Dentist's practice address cannot be confirmed
* The dentist is no longer practicing as of the day before the beginning of the intervention period (December 1, 2023).
* The study team discovers after the time of randomization that dentists are either non-English speaking or have a medical or psychiatric condition that preclude participation in this project (in the judgment of the study team).
* The study team discovers after the time of randomization that the dentist moved to a practice location different from the one had at the time of randomization at any point between the time of randomization and the end of the study period in November 30, 2024. Practice location changes will be assessed based on IQVIA OneKey data as of November 2024. Additionally, the study team will call all included practices up to 2 times during November 2024 to confirm whether the dentist is still practicing at the location.
* The study team discovers after the time of randomization that the dentist stopped practicing dentistry between the time of randomization and the end of the study period on November 30, 2024 (e.g., retirement, death, etc.). This will be assessed using IQVIA (Longitudinal Prescription Database) OneKey data as of November 2024 and by calling practices in November 2024. Additionally, the study team will use 2024 IQVIA data to assess the number of dispensed antibiotic prescriptions in the post-intervention period across all age groups. If this number is zero, this might strongly suggest that the dentist is no longer practicing, as antibiotics are one of the most commonly prescribed classes of medications by dentists.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Differential change in the number of dispensed opioid prescriptions to patients aged 13-30 years between the 8 months before and 8 months after the academic detailing intervention period ends among treatment versus control dentists | 20 months (8 months prior, 4 months for detailing, 8 months after detailing)

SECONDARY OUTCOMES:
Differential change in total morphine milligram equivalents (MMEs) dispensed to patients aged 13-30 years the 8 months before and 8 months after the academic detailing intervention period ends among treatment versus control dentists | 20 months (8 months prior, 4 months for detailing, 8 months after detailing)
Differential change in the number of opioid prescriptions dispensed to patients aged 31 years or older between the 8 months before and 8 months after the academic detailing intervention period ends among treatment versus control dentists | 20 months (8 months prior, 4 months for detailing, 8 months after detailing)
Percentage of participants that complete the initial academic detailing session | 4 months (intervention period)
Satisfaction with the detailing intervention as measured by a follow-up survey on a 5-point Likert scale | Up to three weeks following the academic detailing
  This is a one question survey that participants select from 5 responses: very dissatisfied (1), somewhat dissatisfied (2), neither satisfied nor dissatisfied (3), somewhat satisfied (4), satisfied (5).
Participants willingness to change opioid prescribing practices based on the academic detailing intervention as measured by the follow-up survey on a 5-point Likert scale | Up to three weeks following the academic detailing
  Participants answer one question as to how likely participants will reduce opioid prescribing to adolescents and young adults. The five responses include: very unlikely (1), unlikely (2), neither likely nor unlikely (3), likely (4), very likely (5).

CONTACTS AND LOCATIONS:
Overall Officials: Chad Brummet, M.D., Principal Investigator — University of Michigan; Kao-Ping Chua, MD, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No